CLINICAL TRIAL: NCT04872933
Title: Multicentre Prospective Single-blind Wait-list Randomised Controlled Trial, With Nested Pilot, of the Clinical Value and Economic Evaluation of an Online Physical and Emotional Wellbeing Resource for the Improvement of Health-related Quality of Life in People With Chronic Kidney Disease: The Kidney Beam Trial
Brief Title: The Kidney BEAM Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Bangor University (Other); University of Portsmouth (Other); University of Leicester (Other); Manchester University NHS Foundation Trust (Other Government); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: KCH21-043
Record Dates: First submitted 2021-04-23; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Waitlist (Other): Patient will attend a total of 3 virtual assessments whilst in the study: at baseline, at 12 weeks then at 6 months. The online intervention will commence straight after completing the baseline visit.
  Interventions: Other: Kidney Beam Online Platform
- Waitlist (Other): Patient will be complete assessments at baseline and 12 weeks but will only start the online intervention after the 12-week assessment.
  Interventions: Other: Kidney Beam Online Platform

INTERVENTIONS:
Other: Kidney Beam Online Platform — Kidney Beam is a wellbeing digital health intervention platform that offers patients living with kidney disease a way to improve their physical activity and boost their mental health through live and on demand movement classes and expert educational videos, while remaining in their own home. Kidney Beam is led by specialist kidney professionals, including renal physiotherapists and renal counsellors, from a number of different NHS Trusts and backgrounds, as well as people living with kidney disease.

SUMMARY:
This is a multi-centre single-blind waitlist randomised controlled trial (RCT) that will examine the clinical value and cost-effectiveness of an online physical and emotional wellbeing resource for the improvement of health-related quality of life in people with CKD.

Physical inactivity and poor mental health are very real concerns for people living with kidney disease, and they report multiple symptoms that impact upon the physical component of health-related quality of life (HRQoL). A decrease in the physical component of HRQoL is independently associated with mortality and morbidity. In people living with end stage kidney disease (ESKD), systematic reviews indicate that a range of exercise training interventions improve physical function and alleviate disability symptoms. The physical component of HRQoL can be targeted with interventions to enhance physical activity, however people living with kidney disease are still not routinely offered specialist physical activity or mental health support in the NHS. Kidney Beam is a new wellbeing digital health intervention platform that was developed, and launched, to help people with kidney disease manage their physical and mental health through the Coronavirus 2019 (COVID-19) pandemic, resulting lockdown and beyond. It involves a digital health intervention platform to support people with health conditions to stay physically active. Patients will have access to live-on demand or recorded physical activity classes that they will use for 12 weeks with 2 sessions per week.

The study aims to recruit 304 patients.

DETAILED DESCRIPTION:
Trial Design An investigator-led multicentre single-blind waitlist randomised controlled trial (with nested pilot study) of participants with established chronic kidney disease (CKD). The study will adopt a nested pilot design to preliminarily assess trial and intervention feasibility. To assess this, a traffic light system will be utilised to determine if the study should be halted (red), changes to the design or intervention considered (amber) or is considered feasible and progress to the full trial (green). These criteria will be reviewed and set by the investigators prior to start of study.

Selection of Participants and Procedure

Three hundred and thirty patients aged 18 years or over with established CKD will be enrolled. Potential study trial patients will be identified in outpatient clinic list or approached during their routine hospital visit for an informal chat.

The study team and PI will confirm patient's eligibility. When patient agrees to participate, patient will be asked to sign a consent form. Patient will be scheduled for baseline visit and will be randomised using a secure web-based service. Only by the unblinded member of the study team will be able to randomise patient. Blinded member of the team (research Assistant) will perform the assessment of outcome measures at Baseline and 12 week visit.

After randomisation, patient will be assigned either to waiting list or non-waiting list. If patient is assigned to nonwaiting list group, patient will be asked to attend a total of 3 virtual assessments (baseline, 6M and 12M) and will offered online Kidney BEAM intervention straight away for 12 weeks. If patient is assigned to waiting list group, they will still be asked to complete the 3 virtual assessments but will only start online Kidney BEAM intervention after 12 weeks of being on study. Baseline and 12 week visit will include a review of patient's up to date blood test results, functional capacity (Sit-to stand 60), completion of questionnaire sets and adverse event assessment. After completing the intervention, a highly trained physiotherapist will also conduct qualitative interview to explore patient's experience of the study. For the pilot interviews , up to 15 participants from the intervention arm will be recruited. For the final interviews, up to 30 participants will be recruited in total, from each arm of the trial. Again, data collection will cease at the point where information power is achieved. Interviews are expected to last approximately 60 minutes. At the end of each interview, participants will be given another opportunity to ask questions, or seek clarification and the voluntary nature of their participation will be re-iterated. Should any participant request further information or highlight any concerns during the interview then these will be discussed with the Principal Investigator at their recruiting site, for appropriate onward referral as required.

COVID-19 Sub-study The Kidney Beam trial will contain an exploratory sub-study for any patients with CKD who had COVID-19 or who have been left with CKD following AKI-related to COVID-19 infection. Only patients with history of COVID prior to consent will be assessed using COVID functional status tool at baseline and 12 week visit. Patients who develop COVID while on study will be assessed the same tool on their follow up visit.

For those who had a positive test, an assessment of the severity of their COVID will be made in the following way:

* COVID positive, managed at home not requiring hospital admission
* COVID positive, required hospital admission but no oxygen therapy
* COVID positive, required hospital admission and oxygen therapy
* COVID positive, required hospital admission and non-invasive ventilation
* COVID positive, required hospital admission and admission to intensive care Additional details of the admission, including length of stay and time since discharge will be recorded. Subjects will continue in the study in the same way but will complete the post-COVID functional status tool questionnaire at baseline and follow-up in addition to other outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with established CKD
* Adults aged 18yrs+
* Written or virtual informed consent

Exclusion Criteria:

* Weight < 50kg
* Self-reported participation in a structured exercise programme or kidney beam digital health intervention platform within previous 3 months
* Active infection
* Uncontrolled arrhythmias
* Unstable angina or heart attack within the 3 months
* Persistent uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg)
* Recent (within the last 3 months) stroke or transient ischaemic attack
* Receiving palliative care for advanced terminal cancer
* Patients with peripheral vascular or musculoskeletal disease, who the investigator deems unable to carry out a physical activity intervention.
* Any other health condition considered by the local Principal Investigator in which exercise therapy will be contraindicated.
* Insufficient understanding of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Mental Composite Score (MCS) of KDQOL-36 quality of life questionnaire at 12 weeks. | Week 12
  To assess the clinical value of the Kidney Beam digital health intervention platform

SECONDARY OUTCOMES:
Patient activation measure (PAM-13) | Week 12
  The PAM-13 is a validated tool of 13 questions which assesses a patient's knowledge, skills and confidence in managing their own health.
Chalder Fatigue Questionnaire -- physical and mental fatigue | Baseline and week 12
  The Chalder Fatigue Questionnaire is an 11-item questionnaire measuring the severity of physical and mental fatigue on two separate subscales
Patient Health Questionnaire-4 (PHQ-4) | Baseline
  The Patient-Health Questionnaire-4 (PHQ-4) is an ultra-brief screener for depression and anxiety
Functional capacity | Baseline and Week12
  STS60 (Sit-to-Stand 60 second) to provide a measure of muscle endurance, another aspect of physical performance
Quality of life score | Baseline, Week12 and 6 month follow up
  To assess the quality of life of patients with kidney disease using KDQOL-36 physical component score (PCS), energy/fatigue, burden of kidney disease, role physical, physical functioning, mental health, bodily pain, role emotional, social functioning, general health)
Global Physical Activity Questionnaire | Baseline and Week 12
  It collects information on physical activity participation in three settings (or domains) as well as sedentary behaviour, comprising 16 questions (P1-P16). The domains are:
  * Activity at work
  * Travel to and from places
  * Recreational activities
  It collects information on physical activity participation in three settings (or domains) as well as sedentary behaviour, comprising 16 questions (P1-P16). The domains are:
  * Activity at work
  * Travel to and from places
  * Recreational activities
Clinical Frailty Score | Baseline and Week 12
  The Clinical Frailty Scale (CFS), a risk stratification tool which grades frailty level from 1 (very fit) to 9 (terminally ill) using the standardised qualifiers, and has been validated for use in a range of CKD populations, will be used to identify the frailty status of participants at baseline
Qualitative exploration of intervention and trial acceptability and participant experience | End of 12 week pilot phase and Week 12
  Semi-structured interviews will be used to gather qualitative data as they offer an open and flexible method for exploring the participants' individual experiences in-depth.
Adverse events | Baseline and Week 12
  Episodes of hospitalisation and other infection episodes will be documented and analysed descriptively.
Kidney Beam platform metrics | Week 12
  To assess physical activity and engagement on the Kidney BEAM platform

CONTACTS AND LOCATIONS:
Overall Officials: Sharlene Greenwood, Dr, Principal Investigator — Kings College Hospital NHS Trust
Locations (1):
- Kings College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Greenwood SA, Briggs J, Walklin C, Mangahis E, Young HML, Castle EM, Billany RE, Asgari E, Bhandari S, Bishop N, Bramham K, Burton JO, Campbell J, Chilcot J, Cooper N, Deelchand V, Graham-Brown MPM, Haggis L, Hamilton A, Jesky M, Kalra PA, Koufaki P, McCafferty K, Nixon AC, Noble H, Saynor ZL, Taal MW, Tollitt J, Wheeler DC, Wilkinson TJ, Worboys H, Macdonald J. Kidney Beam-A Cost-Effective Digital Intervention to Improve Mental Health. Kidney Int Rep. 2024 Sep 2;9(11):3204-3217. doi: 10.1016/j.ekir.2024.08.030. eCollection 2024 Nov. PMID 39534205
- [Derived] Young HML, Castle EM, Briggs J, Walklin C, Billany RE, Asgari E, Bhandari S, Bishop N, Bramham K, Burton JO, Campbell J, Chilcot J, Cooper N, Deelchand V, Graham-Brown MPM, Haggis L, Hamilton A, Jesky M, Kalra PA, Koufaki P, Macdonald J, McCafferty K, Nixon AC, Noble H, Saynor ZL, Taal MW, Tollitt J, Wheeler DC, Wilkinson TJ, Greenwood SA. The development and internal pilot trial of a digital physical activity and emotional well-being intervention (Kidney BEAM) for people with chronic kidney disease. Sci Rep. 2024 Jan 6;14(1):700. doi: 10.1038/s41598-023-50507-4. PMID 38184737
- [Derived] Greenwood SA, Young HML, Briggs J, Castle EM, Walklin C, Haggis L, Balkin C, Asgari E, Bhandari S, Burton JO, Billany RE, Bishop NC, Bramham K, Campbell J, Chilcot J, Cooper NJ, Deelchand V, Graham-Brown MPM, Hamilton A, Jesky M, Kalra PA, Koufaki P, McCafferty K, Nixon AC, Noble H, Saynor Z, Taal MW, Tollit J, Wheeler DC, Wilkinson TJ, Worboys H, Macdonald JH. Evaluating the effect of a digital health intervention to enhance physical activity in people with chronic kidney disease (Kidney BEAM): a multicentre, randomised controlled trial in the UK. Lancet Digit Health. 2024 Jan;6(1):e23-e32. doi: 10.1016/S2589-7500(23)00204-2. Epub 2023 Nov 14. PMID 37968170
- [Derived] Walklin CG, Young HML, Asghari E, Bhandari S, Billany RE, Bishop N, Bramham K, Briggs J, Burton JO, Campbell J, Castle EM, Chilcot J, Cooper N, Deelchand V, Graham-Brown MPM, Hamilton A, Jesky M, Kalra PA, Koufaki P, McCafferty K, Nixon AC, Noble H, Saynor ZL, Sothinathan C, Taal MW, Tollitt J, Wheeler DC, Wilkinson TJ, Macdonald JH, Greenwood SA. The effect of a novel, digital physical activity and emotional well-being intervention on health-related quality of life in people with chronic kidney disease: trial design and baseline data from a multicentre prospective, wait-list randomised controlled trial (kidney BEAM). BMC Nephrol. 2023 May 2;24(1):122. doi: 10.1186/s12882-023-03173-7. PMID 37131125